CLINICAL TRIAL: NCT01747876
Title: A Phase I, Multi-center, Open-label Study of LEE011 in Patients With Malignant Rhabdoid Tumors and Neuroblastoma
Brief Title: Study of Safety and Efficacy in Patients With Malignant Rhabdoid Tumors (MRT) and Neuroblastoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of efficacy caused enrollment to be stopped at the end of dose escalation
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLEE011X2102; 2012-004228-40 (EudraCT Number)
Record Dates: First submitted 2012-12-06; First posted 2012-12-12 (Estimated); Results first posted 2019-02-28 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Malignant Rhabdoid Tumors (MRT); Neuroblastoma
Keywords: LEE011; Phase 1; pediatric; CDK4/6 inhibitor; dose escalation; malignant rhabdoid tumors; MRT; neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LEE011 (Experimental)
  Interventions: Drug: LEE011

INTERVENTIONS:
Drug: LEE011 — LEE011 is a small molecule inhibitor of CDK4/6.

SUMMARY:
LEE011 is a small molecule inhibitor of CDK4/6. LEE011 has demonstrated in vitro and in vivo activity in both tumor models. The primary purpose of this study was to determine the maximum tolerated dose (MTD) and/or recommended dose for expansion (RDE) in pediatric patients and to delineate a clinical dose to be used in future studies. This study was also to have assessed the safety, tolerability, PK and preliminary evidence of antitumor activity of LEE011 in patients with MRT or neuroblastoma.

DETAILED DESCRIPTION:
Due to lack of efficacy, enrollment in the study was stopped at the end of dose escalation (sites were notified of the early enrollment halt on 7-Aug-2014) and the dose-expansion part was not conducted. Due to halted enrollment and/or lack of complete responses (CR) and partial responses (PR), efficacy analysis was only performed in terms of TTP for the patients treated during the dose-escalation part at the maximum tolerated dose (MTD) and recommended dose expansion (RDE).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of MRT or, neuroblastoma or in dose escalation part, other tumors with documented evidence of D-cyclin-CDK4/6-INK4a-Rb pathway abnormalities (dose escalation part only),
* Patients with CNS disease should be on stable doses of steroids for at least 7 days prior to first dose of LEE011 with no plans for escalation.
* In expansion part, patients must have at least one measurable disease as defined by RECIST v1.1.
* Patients must have a Lansky (≤ 16 years) or Karnofsky (> 16 years) score of at least 50.

Exclusion Criteria:

* Prior history of QTc prolongation or QTcF > 450 ms on screening ECG.
* Patients with the following laboratory values during screening:

  * Serum creatinine > 1.5 x upper limit of normal (ULN) for age
  * Total bilirubin >1.5 x ULN for age
  * Alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT) > 3 x ULN for age; aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase(SGOT) > 3 x ULN for age except in patients with tumor involvement of the liver who must have AST/SGOT and ALT/SGPT ≤ 5 x ULN for age. For the purpose of this study, the ULN for SGPT/ALT is 45 U/L.
* Patients who are currently receiving treatment with agents that are metabolized predominantly through CYP3A4/5 and have a narrow therapeutic window and/or agents that are known strong inducers or inhibitors CYP3A4/5 are prohibited. In particular, enzyme-inducing antiepileptic drugs (EIAEDs).
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for the study.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2013-05-28 (Actual); Primary Completion 2017-06-29 (Actual); Study Completion 2017-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- United States (6):
  - UCSF Medical Center Dept of Pediatic Oncology, San Francisco, California
  - Childrens Healthcare of Atlanta Dept of Oncology, Atlanta, Georgia
  - Dana Farber Cancer Institute SC-7, Boston, Massachusetts
  - Memorial Sloan Kettering Dept of Onc, New York, New York
  - Cincinnati Children's Hospital Medical Center Dept of Oncology, Cincinnati, Ohio
  - St Jude s Childrens Research Hospital Dept of Oncology, Memphis, Tennessee
- Novartis Investigative Site, Perth, Western Australia, Australia
- France (3):
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Villejuif
- Germany (2):
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Augsburg
- Novartis Investigative Site, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 64 patients were to be treated during the entire study; however, 32 patients were enrolled and treated at the time of the enrollment halt.
Pre-assignment Details: The escalation part of the study explored the 3 doses 280, 350 & 470 mg/m2) in successive cohorts. The dose expansion phase of the study was not conducted (due to enrollment halt).
Groups:
- LEE011 280 mg/m2 - Dose Escalation Only: Patients who took 280 mg/m2 of LEE011
- LEE011 350 mg/m2 - Dose Escalation Only: Patients who took 350 mg/m2 of LEE011. The dose escalation part of the study
- LEE011 470 mg/m2 - Dose Escalation Only: Patients who took 470 mg/m2 of LEE011
Period: Overall Study
Arm/Group | LEE011 280 mg/m2 - Dose Escalation Only | LEE011 350 mg/m2 - Dose Escalation Only | LEE011 470 mg/m2 - Dose Escalation Only
Started | 5 | 15 | 12
Completed | 0 | 0 | 0
Not Completed | 5 | 15 | 12
Not completed — Adverse Event | 1 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Disease progression | 4 | 13 | 8
Not completed — Trtment duration compl. as per protocol | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all patients who received at least one dose of LEE011.
Groups:
- Total: Total of all reporting groups
Arm/Group | LEE011 280 mg/m2 - Dose Escalation Only | LEE011 350 mg/m2 - Dose Escalation Only | LEE011 470 mg/m2 - Dose Escalation Only | Total
Number analyzed (Participants) | 5 | 15 | 12 | 32
Age, Customized [Count of Participants; unit: Participants]
  1 to <2 | 2 | 0 | 1 | 3
  2 to <5 | 2 | 7 | 4 | 13
  6 to <12 | 0 | 3 | 3 | 6
  12 to <18 | 1 | 4 | 2 | 7
  >= 18 | 0 | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 4 | 11
  Male | 4 | 9 | 8 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 2 | 10 | 9 | 21
  Asian | 1 | 0 | 0 | 1
  Other | 0 | 2 | 2 | 4
  Not Available | 2 | 3 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Dose Limiting Toxicities (DLTs) by Primary System Organ Class, Preferred Term and Treatment
Description: A DLT was defined as an AE or clinically significant abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurred within the first 28 days of treatment with LEE011 and met any of the predefined criteria. For the purpose of dose-escalation decisions, DLTs were considered and included in the Bayesian Logistic Regression Model (BLRM). Patients who did not experience DLT during the first cycle were considered to have had sufficient safety evaluations if they were observed for ≥ 28 days following the first dose and were considered to have had enough safety data to conclude that a DLT did not occur. Patients who did not meet these minimum safety evaluation requirements were regarded as ineligible for the DDS. A patient with multiple DLTs within a primary system organ class is counted only once in the total row.
Time Frame: cycle 1 = 28 days (from the time of first dose)
Population: Dose-determining analysis set consisted of all pts from safety set who either met the following minimum exposure criterion & had scheduled safety evaluations, or experienced a DLT. A patient was considered to have met the minimum exposure criterion if he/she had received at least 16 of 21 planned daily doses of LEE011 in first 28 days of dosing.
Measure: Number; unit: Participants
Arm/Group | LEE011 280 mg/m2 - Dose Escalation Only | LEE011 350 mg/m2 - Dose Escalation Only | LEE011 470 mg/m2 - Dose Escalation Only
Number analyzed (Participants) | 5 | 15 | 10
Participants
  Any primary system organ class total | 1 | 0 | 2
  Blood & lymphatic sys. disorders(Thrombocytopenia) | 0 | 0 | 1
  Gen. disorders & admin. site conditions (fatigue) | 1 | 0 | 0
  Investigations (Platelet count decreased) | 0 | 0 | 1

2. Secondary Outcome: Overall Response Rate
Description: This analysis was not done as there were no responders.
Time Frame: Every 2 cycles (cycle = 28 days) up to end of treatment, the maximum time a patient was on study was 1311 days
Population: Full analysis set (FAS) included all patients who received at least one dose of LEE011. This analysis was not done as there were no responders.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | LEE011 280 mg/m2 - Dose Escalation Only | LEE011 350 mg/m2 - Dose Escalation Only | LEE011 470 mg/m2 - Dose Escalation Only
Number analyzed (Participants) | 5 | 15 | 12
months | NA [NA to NA] — This analysis was not done as there were no responders. | NA [NA to NA] — This analysis was not done as there were no responders. | NA [NA to NA] — This analysis was not done as there were no responders.

3. Secondary Outcome: Time to Disease Progression (TTP) Per RECIST 1.1
Description: TTP was assessed per Investigator, for the malignant rhabdoid tumor (MRT) & neuroblastoma patients for the pooled maximum tolerated dose (MTD) & recommended dose for expansion (RDE) according to RECIST 1.1 criteria using Kaplan-Meier method. Time to progression (TTP) is the time from date of randomization/start of treatment to the date of event defined as the first documented progression or death due to underlying cancer. If a patient had not had an event, time to progression was censored at the date of last adequate tumor assessment. At least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Every 2 cycles (cycle = 28 days) up to end of treatment, the maximum time a patient was on study was 1311 days
Population: Full analysis set (FAS) included all patients who received at least one dose of LEE011.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- MRT Group: Patients had a confirmed diagnosis of malignant rhabdoid tumors
- Neuroblastoma (NB): Patients had a confirmed diagnosis of neuroblastoma.
Arm/Group | MRT Group | Neuroblastoma (NB)
Number analyzed (Participants) | 11 | 14
months | 1.8 [1.7 to 2.0] | 1.8 [1.7 to 4.4]

4. Secondary Outcome: Duration of Response (DOR)
Description: Assess the anti-tumor activity of LEE011 by RECIST 1.1. DOR was not assessed.
Time Frame: Every 2 cycles (cycle = 28 days) up to end of treatment, the maximum time a patient was on study was 1311 days
Population: Full analysis set included all patients who received at least 1 dose of LEE011. Due to halted enrollment and/or lack of complete responses (CR) & partial responses (PR), efficacy analysis was only performed in terms of DOR for the patients treated during the dose-escalation part at the MTD and RDE. Therefore, Duration of response was not assessed.
Arm/Group | LEE011 280 mg/m2 - Dose Escalation Only | LEE011 350 mg/m2 - Dose Escalation Only | LEE011 470 mg/m2 - Dose Escalation Only
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Pharmacokinetics (PK) Parameter: AUC0-24
Description: The AUC calculated to the end of a dosing interval (tau) following single dose or at steady-state (amount x time x volume-1). PK parameters were estimated from individual plasma concentration-time profiles using noncompartmental methods in Phoenix WinNonlin.
Time Frame: 0,1, 2, 4, 8 hours post dose Cycle 1 Day 1 (C1D1) and Cycle 1 Day 15 (C1D15)
Population: The pharmacokinetic analysis set (PAS) consisted of all patients who had at least one blood sample providing evaluable drug concentration data.
Measure: Median (Full Range); unit: h*ng/ml
Arm/Group | LEE011 280 mg/m2 - Dose Escalation Only | LEE011 350 mg/m2 - Dose Escalation Only | LEE011 470 mg/m2 - Dose Escalation Only
Number analyzed (Participants) | 5 | 12 | 7
h*ng/ml
  C1D1 | 9250 [4580 to 22000] | 10000 [5320 to 43600] | 17600 [8010 to 28500]
  C1D15: number analyzed (Participants) | 3 | 7 | 5
  C1D15 | 13800 [8910 to 60100] | 24500 [15100 to 60100] | 29100 [13300 to 50500]

6. Secondary Outcome: Pharmacokinetics (PK) Parameter: Cmax
Description: Cmax is the maximum (peak) observed plasma, blood, serum, or other body fluid drug concentration after single dose administration or at steady-state (mass x volume-1). PK parameters were estimated from individual plasma concentration-time profiles using noncompartmental methods in Phoenix WinNonlin
Time Frame: C1D1, C1D15
Population: as for outcome 5
Measure: Median (Full Range); unit: ng/ml
Arm/Group | LEE011 280 mg/m2 - Dose Escalation Only | LEE011 350 mg/m2 - Dose Escalation Only | LEE011 470 mg/m2 - Dose Escalation Only
Number analyzed (Participants) | 5 | 12 | 10
ng/ml
  C1D1: number analyzed (Participants) | 5 | 12 | 7
  C1D1 | 937 [542 to 1910] | 1130 [514 to 4140] | 1960 [796 to 4360]
  C1D15: number analyzed (Participants) | 4 | 12 | 10
  C1D15 | 1110 [860 to 5210] | 2010 [633 to 4270] | 2500 [562 to 5050]

7. Secondary Outcome: Pharmacokinetics (PK) Parameter: Tmax
Description: Tmax is the time to reach maximum (peak) plasma, blood, serum, or other body fluid drug concentration after single dose administration or at steady-state (time). PK parameters were estimated from individual plasma concentration-time profiles using noncompartmental methods in Phoenix WinNonlin.
Time Frame: C1D1, C1D15
Population: as for outcome 5
Measure: Median (Full Range); unit: hour
Arm/Group | LEE011 280 mg/m2 - Dose Escalation Only | LEE011 350 mg/m2 - Dose Escalation Only | LEE011 470 mg/m2 - Dose Escalation Only
Number analyzed (Participants) | 5 | 12 | 10
hour
  C1D1: number analyzed (Participants) | 5 | 12 | 7
  C1D1 | 2.03 [1.1 to 4.08] | 2.02 [1 to 4.05] | 4 [2 to 4.07]
  C1D15: number analyzed (Participants) | 4 | 12 | 10
  C1D15 | 2.08 [1.13 to 3.83] | 2.13 [1.08 to 23.8] | 3.92 [1.98 to 23.6]

ADVERSE EVENTS:
Time Frame: From date of first administration of study treatment to 30 days after date of last actual administration of study
Groups:
- All Patients: All patients who took either 280 mg/m2 or 350 mg/m2 or 470 mg/m2 of LEE011
Arm/Group | LEE011 280 mg/m2 - Dose Escalation Only | LEE011 350 mg/m2 - Dose Escalation Only | LEE011 470 mg/m2 - Dose Escalation Only | All Patients
All-Cause Mortality (participants affected / at risk) | 2/5 | 2/15 | 1/12 | 5/32
Serious Adverse Events (participants affected / at risk) | 3/5 | 7/15 | 4/12 | 14/32
Other Adverse Events (participants affected / at risk) | 5/5 | 15/15 | 12/12 | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LEE011 280 mg/m2 - Dose Escalation Only (N=5) | LEE011 350 mg/m2 - Dose Escalation Only (N=15) | LEE011 470 mg/m2 - Dose Escalation Only (N=12) | All Patients (N=32)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Orbital oedema (Eye disorders) | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Face oedema (General disorders) | 0 | 0 | 1 | 1
Pain (General disorders) | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 2 | 0 | 2
Device related infection (Infections and infestations) | 0 | 1 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 1
Pneumococcal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 1
Pneumococcal infection (Infections and infestations) | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Polydipsia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Central nervous system neuroblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 0 | 1 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1 | 1
Extrapyramidal disorder (Nervous system disorders) | 1 | 0 | 0 | 1
Febrile convulsion (Nervous system disorders) | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 2 | 2
Hydrocephalus (Nervous system disorders) | 0 | 0 | 1 | 1
Intracranial pressure increased (Nervous system disorders) | 1 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 1 | 0 | 1
Irritability (Psychiatric disorders) | 0 | 0 | 1 | 1
Polyuria (Renal and urinary disorders) | 1 | 0 | 0 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LEE011 280 mg/m2 - Dose Escalation Only (N=5) | LEE011 350 mg/m2 - Dose Escalation Only (N=15) | LEE011 470 mg/m2 - Dose Escalation Only (N=12) | All Patients (N=32)
Anaemia (Blood and lymphatic system disorders) | 1 | 8 | 6 | 15
Haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 2 | 3 | 3 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 3 | 4
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 1 | 1 | 3
Deafness (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
External ear inflammation (Ear and labyrinth disorders) | 0 | 1 | 1 | 2
External ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 2 | 0 | 2
Middle ear inflammation (Ear and labyrinth disorders) | 0 | 1 | 1 | 2
Hypothyroidism (Endocrine disorders) | 0 | 1 | 1 | 2
Dry eye (Eye disorders) | 0 | 1 | 0 | 1
Eye discharge (Eye disorders) | 0 | 2 | 0 | 2
Eyelid haematoma (Eye disorders) | 0 | 0 | 1 | 1
Heterophoria (Eye disorders) | 0 | 1 | 0 | 1
Optic atrophy (Eye disorders) | 0 | 1 | 0 | 1
Photophobia (Eye disorders) | 0 | 0 | 1 | 1
Photopsia (Eye disorders) | 0 | 1 | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 1 | 0 | 1
Strabismus (Eye disorders) | 0 | 1 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 5 | 2 | 8
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Anorectal disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 6 | 1 | 7
Diarrhoea (Gastrointestinal disorders) | 3 | 8 | 2 | 13
Dyschezia (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Eructation (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 6 | 5 | 12
Oral disorder (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 2 | 4
Vomiting (Gastrointestinal disorders) | 2 | 12 | 9 | 23
Asthenia (General disorders) | 0 | 5 | 1 | 6
Catheter site pain (General disorders) | 0 | 0 | 1 | 1
Chills (General disorders) | 0 | 1 | 0 | 1
Complication associated with device (General disorders) | 0 | 0 | 1 | 1
Drug intolerance (General disorders) | 0 | 0 | 1 | 1
Face oedema (General disorders) | 0 | 1 | 0 | 1
Fatigue (General disorders) | 1 | 5 | 6 | 12
Gait disturbance (General disorders) | 1 | 1 | 1 | 3
Malaise (General disorders) | 0 | 1 | 1 | 2
Pain (General disorders) | 1 | 1 | 2 | 4
Pyrexia (General disorders) | 1 | 5 | 2 | 8
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 2 | 2 | 5
Device related infection (Infections and infestations) | 0 | 1 | 0 | 1
Foot and mouth disease (Infections and infestations) | 0 | 1 | 0 | 1
Myringitis (Infections and infestations) | 0 | 0 | 1 | 1
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 1
Otitis media (Infections and infestations) | 0 | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 1 | 1
Rash pustular (Infections and infestations) | 0 | 1 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 2 | 2
Skin infection (Infections and infestations) | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 2 | 4
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 4 | 6
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 2
Laceration (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 2
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Scratch (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 3
Alanine aminotransferase increased (Investigations) | 0 | 3 | 2 | 5
Aspartate aminotransferase increased (Investigations) | 0 | 5 | 4 | 9
Bilirubin conjugated increased (Investigations) | 0 | 1 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | 2
Blood bilirubin increased (Investigations) | 0 | 1 | 1 | 2
Blood creatinine decreased (Investigations) | 0 | 1 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 5 | 2 | 7
Blood lactate dehydrogenase decreased (Investigations) | 0 | 1 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 1
Blood potassium decreased (Investigations) | 0 | 1 | 0 | 1
Blood sodium decreased (Investigations) | 0 | 1 | 0 | 1
Blood urea increased (Investigations) | 0 | 1 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 4 | 3 | 7
Gamma-glutamyltransferase increased (Investigations) | 0 | 2 | 0 | 2
Heart rate increased (Investigations) | 0 | 1 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 5 | 5 | 10
Neutrophil count decreased (Investigations) | 0 | 10 | 5 | 15
Platelet count decreased (Investigations) | 0 | 7 | 5 | 12
Weight decreased (Investigations) | 1 | 4 | 1 | 6
Weight increased (Investigations) | 0 | 1 | 1 | 2
White blood cell count decreased (Investigations) | 1 | 11 | 9 | 21
Decreased appetite (Metabolism and nutrition disorders) | 1 | 5 | 2 | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 3
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3 | 0 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 6 | 1 | 8
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 4 | 0 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 5 | 1 | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Bone swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 5 | 2 | 7
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1 | 0 | 1
Brain oedema (Nervous system disorders) | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 2 | 0 | 3
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 1
Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 1 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 3 | 7 | 5 | 15
Hydrocephalus (Nervous system disorders) | 0 | 1 | 0 | 1
IIIrd nerve disorder (Nervous system disorders) | 0 | 1 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 1
Monoplegia (Nervous system disorders) | 1 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 1 | 0 | 2
Syncope (Nervous system disorders) | 0 | 1 | 0 | 1
Tremor (Nervous system disorders) | 0 | 2 | 0 | 2
Aggression (Psychiatric disorders) | 0 | 1 | 0 | 1
Agitation (Psychiatric disorders) | 1 | 2 | 2 | 5
Anxiety (Psychiatric disorders) | 0 | 2 | 0 | 2
Depressed mood (Psychiatric disorders) | 0 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1 | 2 | 4
Irritability (Psychiatric disorders) | 0 | 1 | 0 | 1
Mood altered (Psychiatric disorders) | 2 | 0 | 0 | 2
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Oedema genital (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Bradypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 3 | 9
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 3
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3 | 6
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 4
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2
Rash morbilliform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 0 | 1 | 1 | 2
Hypotension (Vascular disorders) | 0 | 2 | 1 | 3
Raynaud's phenomenon (Vascular disorders) | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2016-02-23): https://cdn.clinicaltrials.gov/large-docs/76/NCT01747876/Prot_000.pdf
  • Statistical Analysis Plan (2016-09-02): https://cdn.clinicaltrials.gov/large-docs/76/NCT01747876/SAP_001.pdf